CLINICAL TRIAL: NCT06279390
Title: Effectiveness of PRE-DELIRIC-Guided SMART/SmART Care in Reducing Delirium Incidence Among Surgical Intensive Care Unit Patients
Brief Title: PRE-DELIRIC Prediction Model Plus SMART Care to Reduce the Incidence of Delirium in ICU Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202305126RINC
Record Dates: First submitted 2023-11-12; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-06

CONDITIONS: Intensive Care Unit Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Delirium is a severe acute brain dysfunction characterised by sudden confusion, inattention and fluctuating level of consciousness, which mainly affects intubated intensive care patients. It increases the risk of self-extubation, prolongs ICU stay and increases mortality. The incidence of delirium in ICUs varies, with approximately 33.3% of patients affected, and rates of new-onset and pre-existing delirium range from 4% to 89%. Accurate diagnosis is challenging, with 60-80% of patients remaining undiagnosed. Early detection is critical for intervention and improved outcomes.

To address these issues, the PREdiction of DELIRium (PRE-DELIRIC) model incorporates 10 risk factors and predicts delirium within 24 hours of ICU admission, allowing risk stratification into low to very high risk categories. It recalibrates predictive values with a sensitivity of 91.3% and specificity of 64.4% using a cut-off score of 27%. However, its integration into delirium management is underexplored. Delirium risk stratification supports efficient resource allocation, cost control, workload reduction and ethical care, while promptly identifying high-risk patients.

In this study, Investigators evaluate the integration of the PRE-DELIRIC model into a comprehensive delirium management approach called PRE-DELIRIC-guided SMART/SmART care. SMART care includes improving familiarity, assessing pain and anxiety, reducing equipment discomfort and cognitive stimulation. Patients with PRE-DELIRIC scores >30% receive SMART care and multidisciplinary involvement, based on the American Delirium Society.

ELIGIBILITY:
Inclusion Criteria:

1. SICU patients are over 18 years old. 2. received surgery intervention

Exclusion Criteria:

1. Clinical diagnosis of mental disorders
2. Underwent neurosurgical procedures,
3. Discharged from the ICU within 24 hours of admission
4. Transitioned to active life support withdrawal or "comfort care only" within 24 hours of ICU admission

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The inclusion criteria encompass patients admitted to a surgical ICU in Taipei, Taiwan, from January 2021 to March 2023.
Sampling Method: Non-Probability Sample
Enrollment: 381 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
the incidence of delirium | duration of ICU stay (postoperative 30 days)
  The incidence of delirium which was assessed by each shift primary ICU nurse by using the ICDSC.

SECONDARY OUTCOMES:
duration of ventilator use | duration of ICU stay( (postoperative 30 days)
  duration of ventilator use
rate of unplanned self-extubation | duration of intubation( (postoperative 30 days)
  indicates the proportion of patients who unintentionally remove their endotracheal tubes (Yes/No)
day of physical restraint | duration of ICU stay (postoperative 30 days)
  day of physical restraint
level of mobility | duration of ICU stay (postoperative 30 days)
  level 0-10 of mobility
cumulative dose of sedatives | duration of ICU stay (postoperative 30 days)
  Sedatives cumulative drugs include midazolam, propofol and dexmedetomidine record 24hours

CONTACTS AND LOCATIONS:
Overall Officials: Wei Ling Hsiao, Master, Principal Investigator — National Taiwan University Hospital; Man-Ling Wang, Doctor, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No